CLINICAL TRIAL: NCT02736292
Title: Mindfulness Practice for Healthcare Professionals in Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20003529
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Stress
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- participant (Experimental)
  Interventions: Behavioral: Mindfulness Practices for Healthcare Professionals

INTERVENTIONS:
Behavioral: Mindfulness Practices for Healthcare Professionals

SUMMARY:
A newly developed intervention, Mindfulness Based Practices for Health Care Professionals in Training: Clinical Applications, will be piloted to determine the feasibility, acceptability, accessibility, and preliminary effects within this population.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professional
* Healthcare professional in training

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Experience of participants regarding feasibility and acceptability | 8 weeks
  open-ended questions (qualitative)

SECONDARY OUTCOMES:
Burnout (MBI) | 8 weeks
  MBI
Perceived stress (PSS) | 8 weeks
  PSS
Depressive symptoms (PHQ9) | 8 weeks
  PHQ9
Mindfulness (FFMQ) | 8 weeks
  FFMQ
Anxiety (STAI) | 8 weeks
  STAI
Ruminations (RRS) | 8 weeks
  RRS

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Kinser, PhD, Principal Investigator — Virginia Commonwealth University

REFERENCES:
- [Derived] Ellen Braun S, Kinser P, Carrico CK, Dow A. Being Mindful: A Long-term Investigation of an Interdisciplinary Course in Mindfulness. Glob Adv Health Med. 2019 Jan 9;8:2164956118820064. doi: 10.1177/2164956118820064. eCollection 2019. PMID 30671283